CLINICAL TRIAL: NCT04885257
Title: A Randomized Placebo-controlled Trial of Methylphenidate in Veterans With a Diagnosis of Post Traumatic Stress Disorder and Recent Cerebral Stroke
Brief Title: Methylphenidate for Ptsd and Stroke Veterans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-011-20F; IK2CX002104 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-13 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: PTSD; Stroke
Keywords: Stress Disorders, Post-Traumatic; stroke
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stroke | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled trial of methylphenidate. One arm receives placebo and the other receives methylphenidate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study personnel and participants will be blinded to the treatment (placebo vs methylphenidate).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patient with both PTSD and recent history of stroke. Placebo control arm. The frequency will be up to twice a day, with oral dosing.
  Interventions: Drug: Placebo
- Methylphenidate (Experimental): Patient with both PTSD and recent history of stroke. Methylphenidate active arm. The oral dosing maximum will be up to 20mg twice daily.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate oral pill. Dosing instructions given to
  Other Names: Concerta, Ritalin
  Arms: Methylphenidate
Drug: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
Veterans with post-traumatic stress disorder (PTSD) have an increased risk of developing ischemic stroke. Veterans enduring PTSD face difficulties in managing their PTSD severity after suffering from a stroke. Currently, clinical trials in PTSD exclude patients with stroke and patients with significant premorbid psychological conditions like PTSD are usually excluded from stroke clinical trials. Methylphenidate (MPH) is a central nervous system stimulant that can improve PTSD symptoms: avoidance behaviors, social withdrawal, hyperarousal, and working memory. MPH can also improve post-stroke outcomes: mood, activities of daily living, and motor functioning. In clinical trials for PTSD or stroke, MPH has been shown to be well-tolerated with minimal adverse events. The high prevalence of PTSD in Veterans with stroke provides strong justification for development of interventions that effectively and simultaneously target both conditions. The overarching goal of our proposal is to understand how MPH improves PTSD severity in Veterans with comorbid stroke.

DETAILED DESCRIPTION:
Veterans with post-traumatic stress disorder (PTSD) have an increased risk of developing ischemic stroke. Veterans enduring PTSD face difficulties in managing their PTSD severity after suffering from a stroke. Currently, clinical trials in PTSD exclude patients with stroke and patients with significant premorbid psychological conditions like PTSD are usually excluded from stroke clinical trials. Methylphenidate (MPH) is a central nervous system stimulant that blocks dopamine and norepinephrine transporters, selectively increasing prefrontal cortex (PFC) activity. MPH can improve PTSD symptoms: avoidance behaviors, social withdrawal, hyperarousal, and working memory. The suspected mechanism is MPH activates PFC, enhancing fear extinction and improving PTSD symptoms. MPH can also improve post-stroke outcomes: mood, activities of daily living, and motor functioning. In clinical trials for PTSD or stroke, MPH has been shown to be well-tolerated with minimal adverse events. The high prevalence of PTSD in Veterans with stroke provides strong justification for development of interventions that effectively and simultaneously target both conditions. The overarching goal of our proposal is to understand how MPH improves PTSD severity in Veterans with comorbid stroke. The purpose of the clinical trial is to evaluate the therapeutic effects on PTSD symptoms and post-stroke recovery of placebo-controlled MPH in Veterans diagnosed with PTSD and cerebral stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veteran of US military; signed informed consent
* Criterion A Index Trauma(s) resulting in PTSD occurred during adulthood prior to stroke
* CAPS-5 past week total score =23 at baseline visit
* Willing to refrain from antipsychotics, mood stabilizers, stimulants, and any formulation of MPH
* First-ever symptomatic ischemic stroke radiologically verified, occurring within past 1-12 months
* Females of child-bearing potential (i.e. not postmenopausal or surgically sterile) must be using a medically acceptable method of birth control and should not be pregnant nor have plans for pregnancy or breastfeeding during the study

Exclusion Criteria:

* Moderate to severe cognitive impairment (Montreal Cognitive Assessment score <16/30)
* Poor pre-stroke baseline function of a modified Rankin score >2
* Presence of any standard MRI contraindications
* Current diagnosis of DSM-5-defined bipolar disorder I, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, or major depressive disorder with psychotic features (MINI)
* Diagnosis of moderate or severe substance use disorder (except for caffeine and nicotine) during the preceding 3 months

  * Patients who utilize alcohol or cannabis but do not meet criteria for moderate or severe disorder are permitted at the discretion of the investigator
  * Participants must agree to abstain from illicit drugs during the study
* Increased risk of suicide that necessitates inpatient treatment or warrants additional therapy excluded by the protocol; and/or intensity of suicidal ideation (Type 4 or Type 5) or any suicidal behavior in the past 3 months on Columbia Suicide Severity Rating Scale (C-SSRS)
* Use of any investigational drug, MPH formulation, antipsychotics, mood stabilizers, monoamine oxidase inhibitors, stimulants or any medication known to be a potent (strong) cytochrome P450 subtype 3A4 inhibitor within 2 weeks of baseline
* Treatment with evidence-based trauma-focused therapy for PTSD within two weeks of baseline (if participant is receiving therapy, he/she must complete treatment prior to entering study)

  * Supportive psychotherapy in process at time of Screening may be continued during the study.
* History of moderate or severe TBI as defined by the Ohio State University TBI Identification Method

  * Based on investigator's clinical judgment, history of mild TBI is not excluded
* Any clinically significant, uncontrolled, or medical/surgical condition or laboratory abnormality that would contraindicate use of MPH (see Human Subjects section)
* Severe allergic reaction, bronchospasm, or hypersensitivity to any MPH formulation.
* Litigating for compensation for a psychiatric disorder. Veterans who are in the process of applying for or receiving VA service-connected disability are eligible
* Current enrollment in another intervention trial for PTSD or stroke
* Persons imprisoned, diagnosed with terminal illness, or require surrogate for consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lin, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAllister TW, Zafonte R, Jain S, Flashman LA, George MS, Grant GA, He F, Lohr JB, Andaluz N, Summerall L, Paulus MP, Raman R, Stein MB. Randomized Placebo-Controlled Trial of Methylphenidate or Galantamine for Persistent Emotional and Cognitive Symptoms Associated with PTSD and/or Traumatic Brain Injury. Neuropsychopharmacology. 2016 Apr;41(5):1191-8. doi: 10.1038/npp.2015.282. Epub 2015 Sep 11. PMID 26361060
- [Background] Grade C, Redford B, Chrostowski J, Toussaint L, Blackwell B. Methylphenidate in early poststroke recovery: a double-blind, placebo-controlled study. Arch Phys Med Rehabil. 1998 Sep;79(9):1047-50. doi: 10.1016/s0003-9993(98)90169-1. PMID 9749682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Methylphenidate
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Methylphenidate | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.30 (11.57) | 65.00 (6.39) | 63.65 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rankin Scale at 12 Weeks
Description: The modified Ranking scale (mRS) is a single-item, global, Likert-type scale ranging from 0-6 (higher scores mean a worse outcome) to categorize level of functional independence with comparison to pre-stroke function, accounting for activities of daily living. Participants were scored at baseline, Week 4, Week 8, Week 12, and 30 days after tapering after methylphenidate/placebo. The mean change from baseline at Week 12 for each group is reported.
Time Frame: From baseline to Week 12
Population: Only participants completing both the baseline and Week 12 mRS assessment were included in this analysis. One participant in the placebo group withdrew before Week 12 so is not included here.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Methylphenidate
Number analyzed (Participants) | 9 | 10
units on a scale | -0.44 (0.53) | -0.50 (1.08)
Statistical Analysis 1: Comparison: Placebo vs Methylphenidate; Test type: Superiority; p = 0.896, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 week study period and the 30 day tapering off methylphenidate/placebo.
Arm/Group | Placebo | Methylphenidate
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10
Other Adverse Events (participants affected / at risk) | 4/10 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Methylphenidate (N=10)
Hospitalization due to infectious illness (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Methylphenidate (N=10)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Speech abnormality (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT04885257/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT04885257/ICF_001.pdf